CLINICAL TRIAL: NCT05119660
Title: Modulation of Frontoparietal Dynamics Underlying Adolescent Working Memory Deficits: A COBRE Pilot Project
Brief Title: Modulation of Frontoparietal Dynamics Underlying Adolescent Working Memory Deficits
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bradley Hospital (Other)
Collaborators: Funding Source: COBRE Center for Neuromodulation at Butler Hospital (Pilot Project) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BradleyH002
Record Dates: First submitted 2021-10-06; First posted 2021-11-15 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2022-10

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Patient Arm (Experimental): In a 2x2 factorial double-blind design, we will randomize a sample of adolescents (13-18 years) with WM deficits to intermittent theta burst stimulation (iTBS) at the left dorsolateral prefrontal cortex (DLPFC) or inferior parietal lobule (IPL), based on each participant's structural brain MRI.
  Participants in both arms will complete an active iTBS session and a sham iTBS session. The primary outcome will be theta-gamma coupling during WM demands, as measured via electroencephalography (EEG) during a Sternberg spatial WM task (SWMT) immediately before and after iTBS.
  Interventions: Device: Intermittent Theta Burst Stimulation
- Healthy Control Arm (Experimental): Control Arm: A sample of healthy young adults (18-25 years) will receive an individualized theta-gamma parameters protocol of iTBS to the left DLPFC.
  Participants in both arms will complete an active iTBS session and a sham iTBS session. The primary outcome will be theta-gamma coupling during WM demands, as measured via electroencephalography (EEG) during a Sternberg spatial WM task (SWMT) immediately before and after iTBS.
  Interventions: Device: Intermittent Theta Burst Stimulation

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation — iTBS

SUMMARY:
The purpose of this study is to test whether a single session of brain stimulation (called repetitive transcranial magnetic stimulation [rTMS]) can improve the brain activity underlying 'working memory.' Working memory is the ability to hold information 'in mind' to complete daily activities. This study involves teenagers with ADHD as well as healthy young adults. It is funded by The COBRE Center for Neuromodulation (CCN) at Butler Hospital (Pilot Project)

DETAILED DESCRIPTION:
The objective of this project is to examine the contributing roles of the PPC and PFC in WM processes and relatedly, develop optimal targets for modulating WM-related neural oscillations. Patient Arm: In a 2x2 factorial double-blind design, we will randomize a sample of adolescents (13-18 years) with WM deficits to intermittent theta burst stimulation (iTBS) at the left dorsolateral prefrontal cortex (DLPFC) or inferior parietal lobule (IPL), based on each participant's structural brain MRI. Control Arm: A sample of healthy young adults (18-25 years) will receive an individualized theta-gamma parameters protocol of iTBS to the left DLPFC. Participants in both arms will complete an active iTBS session and a sham iTBS session. The primary outcome will be theta-gamma coupling during WM demands, as measured via electroencephalography (EEG) during a Sternberg spatial WM task (SWMT) immediately before and after iTBS. The central hypothesis is that the PFC and PPC regions have complimentary roles in executing WM processes. Further, iTBS can modulate theta-gamma coupling in these regions to improve behavioral performance. Our central hypothesis is formulated based on our preliminary data on the critical role of theta-gamma coupling in WM processes. To attain the overall objectives, the following specific aims will be pursued:

Aim 1: Examine the effect of iTBS to the PPC on the encoding stage of WM. Hypothesis: Compared to sham and DLPFC conditions, iTBS to the IPL will increase theta-gamma coupling during encoding. Modulation of theta-gamma coupling will correlate with improved behavioral performance.

Aim 2: Examine the effect of iTBS to the PFC on the maintenance stage of WM. Hypothesis: Compared to sham and IPL conditions, iTBS to the DLPFC will increase theta-gamma coupling during maintenance. Modulation of theta-gamma coupling will correlate with improved behavioral performance.

Aim 3: Examine the feasibility and preliminary effect of individualized iTBS to the PFC. Hypothesis: It will be feasible to utilize peak theta-gamma coupling during the SWMT to identify optimal iTBS parameters. Individualized iTBS will increase theta-gamma coupling during WM demands and improve behavioral performance.

Exploratory Aim: Identify the neocortical circuitry underlying oscillatory modulation. Computational modeling designed for neural interpretation of EEG will translate obtained recordings into cellular/circuit-level activity delineating the neural mechanism of the observed modulation. Hypothesis: pyramidal-interneuron mechanisms within the PPC/PFC will underlie the theta/gamma oscillatory modulation.

ELIGIBILITY:
Patient Arm: We will enroll a sample of adolescents (age 13-18 years) with working memory deficits and ADHD. Participation in this study will not require any adjustments to their clinical care. There are no costs to this study (participants compensated) and there are no expected long-term benefits to the participants. Participants will be compensated for each session. Participants can withdraw from the study at any time.

Inclusion Criteria

1. Ability to provide assent and have parent provide parental permission
2. English fluency of the participant and the legal guardian/parent
3. 13-18 years
4. Parent rating on BRIEF-2 Working Memory: Greater than 1.0 SD above normative mean.
5. IQ > 80
6. Clinical diagnosis of attention deficit hyperactivity disorder (ADHD): predominantly inattentive type, predominantly hyperactive/impulsive type, combined type, or unspecified type. Diagnostic criteria will be confirmed with NICHQ Vanderbilt Assessment Scales-Parent.

Healthy Control Arm: We will target a sample of healthy, young adults. Inclusion Criteria

1. Ability to provide consent
2. English fluency of the participant
3. 18-25 years
4. Never diagnosed or meets current criteria for a psychiatric disorder, as measured by self-report of prior diagnoses and formal completion of the diagnostic interview.

Exclusion Criteria: For patient and healthy control participants

Participants will be screened to exclude individuals with neurological or medical conditions that might confound the results, as well as to exclude participants in whom MRI or TMS might result in increased risk of side effects or complications. Common contraindications include metallic hardware in the body, cardiac pacemaker, patients with an implanted medication pumps or an intracardiac line, or prescription of medications known to lower seizure threshold. These account for the majority of the exclusion criteria listed below:

1. Intracranial pathology from a known genetic disorder (e.g., NF1, tuberous sclerosis) or from acquired neurologic disease (e.g. stroke, tumor), cerebral palsy, history of severe head injury, or significant dysmorphology
2. History of fainting spells of unknown or undetermined etiology that might constitute seizures
3. History of seizures, diagnosis of epilepsy, or immediate (1st degree relative) family history epilepsy
4. Any progressive (e.g., neurodegenerative) neurological disorder
5. Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
6. Contraindicated metal implants in the head, brain or spinal cord (excluding dental implants, braces or fillings)
7. Non-removable makeup or piercings
8. Pacemaker
9. Implanted medication pump
10. Vagal nerve stimulator
11. Deep brain stimulator
12. TENS unit (unless removed completely for the study)
13. Ventriculo-peritoneal shunt
14. Signs of increased intracranial pressure
15. Intracranial lesion (including incidental finding on MRI)
16. History of head injury resulting in prolonged loss of consciousness
17. Substance abuse or dependence within past six months (i.e., DSM-5 substance use disorder criteria)
18. Chronic treatment with prescription medications that decrease cortical seizure threshold, not including psychostimulant medication if deemed to be medically safe as part of the medical review process.
19. Active psychosis or mania
20. Current suicidal intent
21. Current pregnancy
22. Significant visual, hearing or speech impairment
23. Current wards of the state

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in Theta-Gamma Coupling After Sham iTBS | Theta-gamma coupling will be obtained before and after iTBS administration. There will be approximately 5 minutes between the pre and post EEG recordings. The change between pre and post is the outcome variable.
  EEG recording will be obtained while the participant completes the Sternberg Spatial Working Memory Test (SWMT). The coupling between theta phase and gamma amplitude will be extracted from the EEG during encoding and maintaining demands. The change between pre and post a single iTBS session will be calculated.
Change in Theta-Gamma Coupling after Active iTBS | Theta-gamma coupling will be obtained before and after iTBS administration. There will be approximately 5 minutes between the pre and post EEG recordings. The change between pre and post is the outcome variable.
  EEG recording will be obtained while the participant completes the Sternberg Spatial Working Memory Test (SWMT). The coupling between theta phase and gamma amplitude will be extracted from the EEG during encoding and maintaining demands. The change between pre and post a single iTBS session will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- E. P. Bradley Hospital, East Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No